CLINICAL TRIAL: NCT03377023
Title: Phase I/II Study of Nivolumab and Ipilimumab Combined With Nintedanib in Non Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19406
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer, Nonsmall Cell; Non Small Cell Lung Cancer Metastatic
Keywords: Nivolumab; Ipilimumab; Nintedanib; Immunotherapy; Advanced stage non-small cell lung cancer; Locally advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Nintedanib Dose Escalation 100-200 mg QD to BID (Experimental): Nivolumab + Ipilimumab + Nintedanib dose escalation.
  Participants were given the following:
  Nivolumab: 3 mg/kg IV Q2 weeks.
  Ipilimumab: 1 mg/kg Q6 weeks.
  Nintedanib Level -1: 100 mg by mouth (PO) once a day (QD) Days 1-14 (Daily dose =100 mg).
  Nintedanib Level 0:150 mg by mouth (PO) once a day (QD) Days 1-14 (Daily dose =150 mg)
  Nintedanib Level 1: 100 mg PO twice daily (BID) Days 2-28 (Daily dose = 200 mg).
  Nintedanib Level 2: 150 mg PO BID Days 1-14 (Daily dose = 300 mg).
  Nintedanib Level 3: 200 mg PO BID Days 1-14 (Daily dose = 400 mg).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Nintedanib
- Phase 2 - Arm A Nintedanib 100-200 mg BID Treatment-naïve (Active Comparator): Arm A: Treatment-naïve defined as newly diagnosed or treatment-naïve patients, with a target overall response rate (ORR) of 50%.
  Participants were given the following:
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks. Ipilimumab: Intravenous ipilimumab every 6 weeks. Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Nintedanib
- Phase 2 - Arm B Nintedanib 100-200 mg BID Treatment Non-naïve (Active Comparator): Arm B: Treatment Non-naïve defined as patients who have been previously exposed to immunotherapy, such as anti-PD-1, anti-PD-L1 or anti-CTLA-4, with a target ORR of 20%.
  Participants were given the following:
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks. Ipilimumab: Intravenous ipilimumab every 6 weeks. Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Nintedanib

INTERVENTIONS:
Drug: Nivolumab — Intravenous nivolumab every 2 weeks.
  Other Names: Opdivo®
Drug: Ipilimumab — Intravenous ipilimumab every 6 weeks.
  Other Names: Yervoy®
Drug: Nintedanib — Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
  Other Names: Vargatef®; Ofev®; BIBF1120

SUMMARY:
The main purpose of this study is to see if the combination of nivolumab, ipilimumab and nintedanib is effective in people with non- small cell lung cancer. Researchers also want to find out if the combination of nivolumab, ipilimumab and nintedanib is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytological diagnosis of advanced/metastatic Non-Small Cell Lung Cancer (NSCLC) with no curative treatment options. For those with mixed histology, there must be a predominant histology.
* 18 years of age or older on day of signing informed consent.
* Life expectancy of at least 3-6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 and 1
* For phase I trial portion, treatment naïve or patients previously treated with chemotherapy, immunotherapy or targeted therapy for NSCLC are allowed. Patient who underwent curative intent chemotherapy and/radiation in the neoadjuvant or adjuvant setting are allowed to enroll if tumor recurrence occurred greater than 6 months from completion of that therapy (and will be considered treatment naïve in the Stage IV setting). Patients with NSCLC tumor known to harbor a genomic aberration for which FDA approved treatment is available (i.e, non-resistant EGFR mutations, EGFR T790M mutation, ALK rearrangement, ROS rearrangement, BRAF V600E mutation) are allowed to enroll if they have received prior treatment with the FDA approved targeted therapy.
* For phase II trial portion, Patients will be enrolled as two parallel cohorts:

  * A.) Arm A (treatment naïve): Patients who are newly diagnosed and treatment naïve. Patient who underwent curative intent chemotherapy and/radiation in the neoadjuvant or adjuvant setting are allowed to enroll if tumor recurrence occurred greater than 6 months from completion of therapy. Patients with NSCLC tumor known to harbor a genomic aberration for which FDA approved treatment is available (i.e, non-resistant EGFR mutations, EGFR T790M mutation, ALK rearrangement, ROS rearrangement, BRAF V600E mutation) are allowed to enroll if they have received prior treatment with the FDA approved targeted therapy.
  * B.) Arm B (Immunotherapy pre-treated group): Patients who have received prior immunotherapy. Patients who are primary refractory to immunotherapy (i.e., Patients who were previously treated with immunotherapy and did not at least achieve stable disease on first imaging assessment on immunotherapy) or have relapsed disease (i.e., Patients that were treated with immunotherapy, achieved at least stable disease on first imaging assessment and subsequently developed disease progression or relapse). Patients with NSCLC tumor known to harbor a genomic aberration for which FDA approved treatment is available (i.e, non-resistant EGFR mutations, EGFR T790M mutation, ALK rearrangement, ROS rearrangement, BRAF V600E mutation) are allowed to enroll if they have received prior treatment with the FDA approved targeted therapy
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
* QTcB must be <470 ms for males and <480 ms for females.
* Adequate normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >1.5 x 10^9/L (> 1500 per mm^3)
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3)
  * Total bilirubin ≤ 1.5 X normal institutional limits. For patients with liver metastasis: total bilirubin must be within normal limits.
  * Proteinuria less than Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater
  * (Except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL
  * AST (SGOT)/ALT(SGPT) ≤1.5 X institutional upper limit of norma (ULN)l or ≤ 2.5 X ULN for patients with liver metastases. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * Serum creatinine CL ≤ 1.5 X ULN or creatinine clearance > 45 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* Have archival tissue where available.
* In addition, patients enrolled on the clinical trial must be willing and able to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Patients for whom newly obtained samples cannot be provided may submit an archived specimen only upon agreement from the Sponsor.
* Female participants of childbearing potential should have a negative urine or serum pregnancy within 72 hours before receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Ability to understand and willingness to provide written informed consent signed and dated prior to admission to the study in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines and to the local legislation.

Exclusion Criteria:

* Concurrent use of other anticancer agents including chemotherapy, targeted therapy, radiotherapy or immunotherapy not otherwise specified in the protocol.
* Concurrent use of other investigational drugs or treatment in another clinical trial with a non- FDA-approved medication within the past 4 weeks before start of therapy.
* Chemo-, or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 2 weeks prior to treatment with the trial drug.
* Radiotherapy (except for brain and extremities or stereotactic treatment) within the past 2 weeks prior to treatment with the trial drug.
* In immunotherapy pretreated patients, any history of dose-limiting toxicity with prior immunotherapy agents, including grade 3/4 immune-related adverse events (irAEs); irreversible irAEs; Grade ≥3 irAEs that did not respond to steroid rescue; or neurologic irAE with significant clinical sequelae.
* Prior treatment with nintedanib (BIBF1120).
* Known hypersensitivity to nintedanib, nivolumab, ipilimumab, peanut or soy or any other trial drug, or their excipients.
* Any toxicity (>CTCAE version 5 grade 3) from previous anti-cancer therapy that has not resolved to a Grade 1. Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy, alopecia).
* History of leptomeningeal carcinomatosis.
* Radiotherapy to a target lesion within the past 3 months prior to baseline imaging unless that area has demonstrated progression.
* Active brain metastases (e.g., stable for <2 weeks, symptomatic, no adequate previous treatment, requiring treatment with anti-convulsants); dexamethasone therapy will be allowed if administered as stable or decreasing dose for at least 3 weeks before randomization otherwise no steroids to exceed prednisone 10 mg/day prior to starting trial treatment. Symptomatic or uncontrolled central nervous system (CNS) metastasis.
* Current or prior use of immunosuppressive medication 7 days before the first dose of nivolumab or ipilimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. A brief course (≤28 days) of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted. Topical corticosteroids are permitted.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, type I diabetes mellitus or residual hypothyroidism due to autoimmune condition only requiring hormone replacement, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Therapeutic anticoagulation with drugs requiring INR monitoring (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or antiplatelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg per day.
* Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* History of clinically significant hemorrhagic or thromboembolic event in the past 6 months.
* Known inherited predisposition to bleeding or thrombosis.
* Significant cardiovascular diseases (i.e., uncontrolled hypertension, unstable angina, history of infarction within the past 3 months prior to start of study treatment, congestive heart failure > New York Heart Association (NYHA) II, serious cardiac arrhythmia).
* Coagulation parameters: International normalized ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional ULN.
* History of another primary malignancy within the past 2 years except for:

  * Basal cell skin cancer
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ)
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* History of known active primary immunodeficiency
* History of allogeneic organ transplant
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study treatment.
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g., such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) for the duration specified during the trial and after end of active therapy
* Pregnancy or breastfeeding female patients must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment
* Psychological, familial, sociological, or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
* Active alcohol or drug abuse
* Significant weight loss (> 20% of Body Weight) within past 6 months prior to inclusion into the trial
* History of active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle E. Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg); Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg); Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg): Nivolumab + Ipilimumab + Nintedanib Dose Escalation.
  Participants were given a fixed dose of Nivolumab 3 mg/kg IV every 2 weeks, a fixed dose of Ipilimumab 1 mg/kg every 6 weeks, and escalating doses of Nintedanib starting at 100mg PO once daily (five dose levels) to determine the Maximum Tolerated Dose (MTD).
- Phase 2 - Arm A Nintedanib 200 mg BID Treatment-naïve: Arm A: Treatment-naïve defined as newly diagnosed or treatment-naïve patients, with a target overall response rate (ORR) of 50%.
  Participants were given the following:
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks.
  Ipilimumab: Intravenous ipilimumab every 6 weeks.
  Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
- Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve: Arm B: Treatment Non-naïve defined as patients who have been previously exposed to immunotherapy, such as anti-PD-1, anti-PD-L1 or anti-CTLA-4, with a target ORR of 20%.
  Participants were given the following:
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks.
  Ipilimumab: Intravenous ipilimumab every 6 weeks.
  Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
Period: Overall Study
Arm/Group | Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg) | Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg) | Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg) | Phase 2 - Arm A Nintedanib 200 mg BID Treatment-naïve | Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve
Started | 3 | 6 | 5 | 22 | 30
Completed | 3 | 6 | 5 | 22 | 30
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable Participants
Groups:
- Phase 2- Arm A Nintedanib 200 mg BID Treatment-naïve: Arm A: Treatment-naïve defined as newly diagnosed or treatment-naïve patients, with a target overall response rate (ORR) of 50%.
  Participants were given the following:
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks.
  Ipilimumab: Intravenous ipilimumab every 6 weeks.
  Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg) | Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg) | Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg) | Phase 2- Arm A Nintedanib 200 mg BID Treatment-naïve | Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve | Total
Number analyzed (Participants) | 3 | 6 | 5 | 22 | 28 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 9 | 13 | 29
  >=65 years | 2 | 3 | 2 | 13 | 15 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 12 | 15 | 35
  Male | 2 | 3 | 1 | 10 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 2 | 6 | 5 | 20 | 25 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 2 | 3
  White | 3 | 6 | 5 | 20 | 23 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 5 | 22 | 29 | 65

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD)
Description: Dose escalation to determine the MTD and Recommended Phase 2 Dose (RP2D) of concurrent administration of nivolumab, ipilimumab, and nintedanib. The maximum tolerated dose (MTD) is defined as the dose with the dose limiting toxicity (DLT) rate of 30%. Phase 1 began with 100 mg nintedanib, 3 mg/kg IV nivolumab + 1 mg/kg ipilimumab. Dosing of nintedanib increased by 50 mg in each level until dose limiting toxicity.
Time Frame: Up to 12 months
Population: Phase 1 participants
Measure: Number; unit: miligrams nintedanib
Groups:
- Phase 1-Dose Escalation: Nivolumab + Ipilimumab + Nintedanib dose escalation
Arm/Group | Phase 1-Dose Escalation
Number analyzed (Participants) | 14
miligrams nintedanib | 150

2. Primary Outcome: Phase 2 - Objective Response Rate (ORR) Per Treatment Arm
Description: Objective response is defined as confirmed CR or confirmed PR based on modified RECIST guidelines version 1.1. The ORR will be estimated by calculating the proportion of patients who achieve OR; the 80% Confidence Interval (CI) and 95% CI for the OR rate will be estimated using the exact binomial distribution. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2 - Arm A: Arm A: Newly diagnosed or treatment-naïve patients, with a target overall response rate (ORR) of 50%.
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks.
  Ipilimumab: Intravenous ipilimumab every 6 weeks.
  Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
- Phase 2 - Arm B: Arm B: Patients who have been previously exposed to immunotherapy, such as anti-PD-1, anti-PD-L1 or anti-CTLA-4, with a target ORR of 20%.
  Nivolumab + Ipilimumab + Nintedanib at RP2D.
  Nivolumab: Intravenous nivolumab every 2 weeks.
  Ipilimumab: Intravenous ipilimumab every 6 weeks.
  Nintedanib: Nintedanib 100-200 mg capsules by mouth twice daily for two-week cycles.
Arm/Group | Phase 2 - Arm A | Phase 2 - Arm B
Number analyzed (Participants) | 22 | 28
percentage of participants | 40.9 [21.5 to 63.3] | 21.4 [9.03 to 41.5]

3. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: Disease control is defined as CR, PR, or SD based on RECIST guidelines version 1.1 with modifications. The disease control rate (DCR) will be estimated by the proportion of patients who achieve DC, and its 80% CI and 95% CI will be estimated using the exact binomial distribution. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 - Arm A | Phase 2 - Arm B
Number analyzed (Participants) | 22 | 28
percentage of participants | 72.7 [49.6 to 88.4] | 57.1 [37.4 to 75.0]

4. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival will be determined as the time from the start of treatment with nivolumab plus ipilimumab plus nintedanib until death due to any cause. For patients who are alive at the time of data cut-off, OS will be censored on the last date when patients are known to be alive. This result is provided as number of months of survival.
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 - Arm A | Phase 2 - Arm B
Number analyzed (Participants) | 22 | 28
months | 17.1 [5.5 to 46.9] | 8.2 [5.0 to 25.3]

5. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Up to 36 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 - Arm A | Phase 2 - Arm B
Number analyzed (Participants) | 22 | 28
months | 5.5 [2.9 to 36.0] | 2.6 [1.4 to 6.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from start of Study Treatment to 100 days from end of treatment. Approximately 57 Months.
Arm/Group | Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg) | Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg) | Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg) | Phase 2- Arm A Nintedanib 200 mg BID Treatment-naïve | Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/6 | 5/5 | 19/22 | 23/30
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/6 | 4/5 | 14/22 | 15/30
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 22/22 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg) (N=3) | Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg) (N=6) | Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg) (N=5) | Phase 2- Arm A Nintedanib 200 mg BID Treatment-naïve (N=22) | Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve (N=30)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Autoimmune mediated hepatitis (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Nintedanib Level -1: 100 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 100 mg) (N=3) | Phase 1 Nintedanib Level 0: 150 mg by Mouth (PO) Once a Day (QD) Days 1-14 (Daily Dose 150 mg) (N=6) | Phase 1 Nintedanib Level 1: 100 mg by Mouth (PO) Twice Daily (BID) Days 2-28 (Daily Dose 200 mg) (N=5) | Phase 2- Arm A Nintedanib 200 mg BID Treatment-naïve (N=22) | Phase 2- Arm B Nintedanib 200 mg BID Treatment Non-naïve (N=30)
Fatigue (General disorders) | 2 (3) | 6 (6) | 2 (7) | 12 (16) | 16 (19)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (2) | 0 (0) | 7 (8) | 5 (11)
Pain (General disorders) | 1 (2) | 3 (4) | 0 (0) | 6 (6) | 3 (8)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 5 (6)
Edema Limbs (General disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 3 (8)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (6) | 2 (4) | 14 (26) | 16 (30)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 1 (7) | 14 (25) | 12 (26)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 6 (9) | 7 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (8) | 1 (2) | 3 (7) | 9 (15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (12) | 7 (9)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Colitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (4) | 5 (6) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 5 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (6) | 1 (1) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 2 (2) | 9 (12) | 13 (17)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 0 (0) | 3 (8) | 7 (23)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 4 (6) | 1 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (5) | 3 (8) | 4 (10) | 7 (9)
Investigations - Other, specify (Investigations) | 1 (2) | 4 (10) | 3 (3) | 5 (9) | 5 (11)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (7) | 3 (7) | 3 (12) | 7 (11)
Weight loss (Investigations) | 1 (1) | 2 (3) | 1 (1) | 3 (4) | 4 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (4) | 2 (3) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 1 (1) | 2 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (13) | 5 (7)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 6 (11) | 8 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (8) | 2 (4) | 2 (2) | 4 (9)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (14) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Alopecia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Scalp pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 5 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 3 (7) | 2 (8)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (5)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (6)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 4 (6) | 6 (21)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (8)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03377023/Prot_SAP_000.pdf